CLINICAL TRIAL: NCT03627832
Title: Insomnia Treatment and Problems (the iTAP Study)
Acronym: iTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Mary E Miller, Professor, Psychiatry, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010684; DXV15 (Other Grant/Funding Number: University of Missouri Research Board)
Record Dates: First submitted 2018-07-23; First posted 2018-08-13 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Insomnia; Alcohol; Harmful Use
Keywords: alcohol; drinking; sleep; insomnia; young adult
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to receive either Cognitive Behavioral Therapy for Insomnia (CBT-I) or Sleep Hygiene.
Who Masked: Participant, Outcomes Assessor
Masking Description: PI Miller will not be blinded to block size or participant assignment because she will inform study therapists of participant assignment to conditions. However, PI Miller and study therapists will be blinded to assessment outcomes, and the assessment RA will be blinded to participant condition. All participants will be told that they will be assigned to one of two insomnia treatment conditions in order to blind them to condition assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I (Experimental): Individual Cognitive Behavioral Therapy for Insomnia (CBT-I) delivered once a week for 6 weeks
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I); Behavioral: Sleep Hygiene
- Sleep Hygiene (Active Comparator): Sleep hygiene handout delivered once to all participants
  Interventions: Behavioral: Sleep Hygiene

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — Participants assigned to the CBT-I condition will attend 1-hour individual sessions of CBT-I once a week for five weeks. Consistent with clinical guidelines (Schutte-Rodin, Broch, Buysse, Dorsey, & Sateia, 2008), treatment will include stimulus control (e.g., limit use of bed to sleep or sexual activity, get out of bed if lying awake for more than 20 minutes), sleep restriction (limit time in bed to amount of time spent sleeping on a typical night), sleep hygiene (e.g., avoid exercise within 2 hours of bedtime, create cool and dark sleep environment), relaxation training, and cognitive restructuring.
  Arms: CBT-I
Behavioral: Sleep Hygiene — All participants will receive a one-page handout on sleep hygiene. This is the only intervention that participants assigned to the Sleep Hygiene condition will receive and is consistent with what may be expected as standard care in a doctor's visit with a primary care physician.

SUMMARY:
This project aims to evaluate the efficacy of insomnia treatment in improving insomnia symptoms and alcohol-related problems among heavy-drinking young adults.

DETAILED DESCRIPTION:
Heavy alcohol use is prevalent among young adults and results in significant physical and psychological burden. Despite wide implementation of alcohol risk reduction efforts on college campuses, rates of heavy alcohol consumption remain high, with 35% of students reporting consumption of 5+ drinks on the same occasion in the past 2 weeks. Thus, additional strategies are needed to reduce the burden of heavy alcohol use among college students. More than half of heavy-drinking college students report symptoms of insomnia. In turn, insomnia symptoms have been associated with increased risk of alcohol-related problems. The proposed project aims to reduce the burden of heavy alcohol use on college campuses by examining the efficacy of Cognitive Behavioral Therapy for Insomnia (CBT-I) in reducing alcohol use and related problems among heavy-drinking college students. Twenty seven young adults who indicate risk for problem drinking and meet DSM-5 criteria for Insomnia Disorder will participate in a 5-week pilot trial. Participants will complete five individual sessions of CBT-I. Outcomes will be assessed at the end of the active intervention period (6 weeks) and 1 month post-intervention. Outcomes of interest include insomnia severity, total wake time, sleep quality, drinking quantity, and alcohol-related consequences. The proposed research aims to reduce the harms associated with heavy alcohol use among young adults by improving the availability of efficacious treatment. It will impact understanding of the benefits of CBT-I, and it is innovative because it evaluates improvement in insomnia as a mechanism for improvements in alcohol use disorder (AUD). This research is consistent with the National Institute on Alcohol Abuse and Alcoholism's initiative to evaluate and promote interventions that prevent the progression of AUD in diverse populations. It will enhance the stature of the university by improving our ability to compete successfully for federal funding to conduct high-quality research.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years
* Heavy episodic drinking, defined as 1 heavy drinking episode (4/5+ drinks for women/men) in the past 30 days on the Timeline Followback
* DSM-5 criteria for insomnia, with "daytime impairment" operationalized as ISI scores =>10

Exclusion Criteria:

* Unable to provide informed consent
* New sleep medication in the past 6 weeks
* Contraindications for CBT-I (mania or seizure disorder)
* Severe psychiatric disorder that requires clinical attention (PTSD, major depression)
* Current treatment for insomnia or alcohol use

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Miller, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

REFERENCES:
- [Derived] Miller MB, Carpenter RW, Freeman LK, Curtis AF, Yurasek AM, McCrae CS. Cannabis use as a moderator of cognitive behavioral therapy for insomnia. J Clin Sleep Med. 2022 Apr 1;18(4):1047-1054. doi: 10.5664/jcsm.9796. PMID 34870584
- [Derived] Miller MB, Curtis AF, Hall NA, Freeman LK, Everson AT, Martinez LD, Park CJ, McCrae CS. Daily associations between modifiable sleep behaviors and nighttime sleep among young adult drinkers with insomnia. J Clin Sleep Med. 2022 Mar 1;18(3):703-712. doi: 10.5664/jcsm.9706. PMID 34605392
- [Derived] Miller MB, Freeman LK, Deroche CB, Park CJ, Hall NA, McCrae CS. Sleep and alcohol use among young adult drinkers with Insomnia: A daily process model. Addict Behav. 2021 Aug;119:106911. doi: 10.1016/j.addbeh.2021.106911. Epub 2021 Mar 15. PMID 33773200
- [Derived] Miller MB, Deroche CB, Freeman LK, Park CJ, Hall NA, Sahota PK, McCrae CS. Cognitive behavioral therapy for insomnia among young adults who are actively drinking: a randomized pilot trial. Sleep. 2021 Feb 12;44(2):zsaa171. doi: 10.1093/sleep/zsaa171. PMID 32886778

RESULTS

PARTICIPANT FLOW:
Groups:
- CBT-I: Individual Cognitive Behavioral Therapy for Insomnia (CBT-I) delivered once a week.
  Participants will attend 1-hour individual sessions of CBT-I once a week for five weeks. Consistent with clinical guidelines (Schutte-Rodin, Broch, Buysse, Dorsey, & Sateia, 2008), treatment will include stimulus control (e.g., limit use of bed to sleep or sexual activity, get out of bed if lying awake for more than 20 minutes), sleep restriction (limit time in bed to amount of time spent sleeping on a typical night), sleep hygiene (e.g., avoid exercise within 2 hours of bedtime, create cool and dark sleep environment), relaxation training, and cognitive restructuring.
  Participants will also receive a one-page handout on sleep hygiene that is consistent with what may be expected as standard care in a doctor's visit with a primary care physician.
- Sleep Hygiene: Participants will receive a one-page handout on sleep hygiene that is consistent with what may be expected as standard care in a doctor's visit with a primary care physician.
Period: Overall Study
Arm/Group | CBT-I | Sleep Hygiene
Started | 28 | 28
Completed | 18 | 27
Not Completed | 10 | 1
Not completed — Withdrawal by Subject | 10 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-I | Sleep Hygiene | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (2.7) | 22.5 (2.8) | 22.5 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56
Alcohol Use Disorder [Count of Participants; unit: Participants] | 25 | 22 | 47
College Enrollment [Count of Participants; unit: Participants] | 21 | 20 | 41
Comorbid Mental Health Disorder [Count of Participants; unit: Participants] | 14 | 10 | 24
Insomnia Severity [Mean (Standard Deviation); unit: units on a scale] — Insomnia Severity measured using the Insomnia Severity Index. Participants rate how severe their concerns are to seven sleep-related questions on a scale of 0-4, where higher scores indicate worse insomnia. Total scores range from 0-28.
  units on a scale | 16.43 (4.06) | 15.93 (2.92) | 16.04 (4.01)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity
Description: Assessed using the Insomnia Severity Index. Scores range from 0 to 28, with higher scores indicating higher insomnia severity.
Time Frame: Change from baseline to post-treatment (week 8) to 1 month follow-up (week 12)
Measure: Mean (Standard Deviation); unit: units on scale, Insomnia Severity Index
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 28 | 28
units on scale, Insomnia Severity Index
  Post Treatment | 6.86 (3.66) | 10.84 (3.5)
  1-Month Follow-Up | 6.58 (3.41) | 9.32 (4.8)

2. Primary Outcome: Sleep Efficiency
Description: Assessed using daily sleep diaries and actigraphy -- sleep efficiency is the proportion of time spent in bed (from lights out until out of bed in the morning) that is actually spent sleeping (subtracting how long it took to fall asleep and how much time was spent awake in the middle of the night).
Time Frame: Change from baseline to post-treatment (week 8) to 1 month follow-up (week 12)
Measure: Mean (Standard Deviation); unit: % of time spent in bed actually asleep
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 28 | 28
% of time spent in bed actually asleep
  Post Treatment | 79.27 (7.95) | 76.48 (7.09)
  1-Month Follow-Up | 76.22 (9.8) | 76.54 (7.94)

3. Primary Outcome: Sleep Quality
Description: Assessed using a single question on the daily sleep diary. Sleep quality score ranges from 0-4, where 0=very poor sleep quality and 4=very good sleep quality.
Time Frame: Change from baseline to post-treatment (week 8) to 1 month follow-up (week 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 28 | 28
units on a scale
  Post Treatment | 2.25 (.66) | 2.32 (.62)
  1-Month Follow-Up | 2.49 (.62) | 2.29 (.55)

4. Primary Outcome: Drinking Quantity
Description: Assessed using the Daily Drinking Questionnaire. Participants estimate how many alcoholic drinks they typically consume on each day of the week, averaged over the past 3 months.Responses for drinking quantity range from 0 to infinity, where higher numbers indicate more standard drinks consumed per day. Reports from each day are summed to create a "Drinks Per Week" score. Participants also report the amount of time they typically spend drinking during each day of the week. Responses range from 0-24 hours per day, where higher numbers indicate more hours drinking.
Time Frame: Change from baseline to post-treatment (week 8) to 1 month follow-up (week 12)
Measure: Mean (Standard Deviation); unit: Drinks per Week
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 28 | 28
Drinks per Week
  Post Treatment | 11.45 (8.25) | 11.80 (9.20)
  1-Month Follow-Up | 8.7 (7.70) | 9.33 (8.77)

5. Primary Outcome: Alcohol-related Consequences
Description: Assessed using the Brief Young Adult Alcohol Consequences Questionnaire. Scores range from 0-24, with higher scores indicating more alcohol-related consequences.
Time Frame: Change from baseline to post-treatment (week 8) to 1 month follow-up (week 12)
Measure: Mean (Standard Deviation); unit: units on a scale - BYAAC
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 28 | 28
units on a scale - BYAAC
  Post Treatment | 4.18 (5.53) | 5.01 (4.18)
  1-Month Follow-Up | 5.04 (5.15) | 3.47 (3.17)

6. Secondary Outcome: Delay Discounting
Description: Assessed using the Monetary Choice Questionnaire. Responses will be used to calculate discount rate (k), consistency of the discount rate (the inferred k), and the proportion of immediate reward choices (immediate choice ratios).
Time Frame: Change from baseline to post-treatment (week 8) to 1 month follow-up (week 12)
Population: Secondary data have not been analyzed yet.
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Negative Affect
Description: Assessed using the Positive and Negative Affect Schedule. Participants respond to words that describe negative feelings/emotions and report the extent (1-5) that they feel each emotion presently or during the past week. Higher scores indicate higher negative affect.
Time Frame: Change from baseline to post-treatment (week 8) to 1 month follow-up (week 12)
Population: Secondary data have not been analyzed yet.
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Emotion Regulation
Description: Assessed using the Difficulties with Emotion Regulation Scale. Scores range from 36-180, with higher scores indicating more difficulty with emotion regulation.
Time Frame: Change from baseline to post-treatment (week 8) to 1 month follow-up (week 12)
Population: Secondary data not analyzed yet.
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Alcohol Craving
Description: Assessed using the Penn Alcohol Craving Scale. Scores range from 0-30, with higher scores indicating greater alcohol craving.
Time Frame: Change from baseline to post-treatment (week 8) to 1 month follow-up (week 12)
Population: Secondary data not analyzed yet.
Arm/Group | CBT-I | Sleep Hygiene
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 11 Weeks
Arm/Group | CBT-I | Sleep Hygiene
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03627832/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-03-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT03627832/Prot_SAP_001.pdf